CLINICAL TRIAL: NCT02405910
Title: A Phase II Randomized Study of Nab-paclitaxel With Gemcitabine at Two Different Dose Combinations to Determine Efficacy in Patients With Advanced Non- Squamous Non-small Cell Lung Cancer (NSCLC).
Brief Title: Ph2 Nab-paclitaxel With Gemcitabine to Determine Efficacy in Advanced Non-squamous NSCLC.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Left Institution
Sponsor: West Virginia University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WVU020514
Record Dates: First submitted 2015-03-24; First posted 2015-04-01 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: advanced; non-squamous; first line therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - Nab-paclitaxel 100mg + Gemcitabine 1250mg (Experimental): Nab-paclitaxel 100 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) on days 1, 8 and 15 of a 21 day cycle. On days 1 and 8 of each cycle, nab-paclitaxel administration will be followed by the administration of gemcitabine 1250 mg/m2 as a 30 minute infusion (maximum 40 minutes).
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine
- B - Nab-paclitaxel 125mg + Gemcitabine 1000mg (Experimental): Nab-paclitaxel 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) on days 1, 8 and 15 of a 28 day cycle. Each nab-paclitaxel administration will be followed by the administration of gemcitabine 1000 mg/m2 as a 30 minute infusion (maximum 40 minutes) on days 1, 8 and 15. Treatments will be repeated until progression or intolerance.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab-paclitaxel
  Other Names: Abraxane; ABI-007
Drug: Gemcitabine
  Other Names: Gemzar; LY-188011

SUMMARY:
Phase II study to determine progression free survival (PFS) of nab-paclitaxel administered in combination with gemcitabine, at two different dose combinations as first line therapy in patients with unresectable stage IIIB/stage IV non-squamous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This study is designed determine progression free survival (PFS) of nab-paclitaxel administered in combination with gemcitabine at two different dose combinations in patients with unresectable stage IIIB/stage IV non-squamous non-small cell lung cancer (NSCLC). Two dosing strategies of the nab-paclitaxel plus gemcitabine combination will be compared for efficacy and tolerability. One arm will combine both agents at their current Food and Drug Administration (FDA) approved doses for the indication of non-small cell lung cancer (NSCLC). This arm will utilize gemcitabine 1250 mg/m2 IV day 1 and day 8 (FDA approved dose in combination with cisplatin) combined with nab-paclitaxel 100 mg/m2 IV day 1, 8 and 15 every 21 days (FDA approved dose in combination with carboplatin). The second arm will utilize the drugs at doses that are approved by the FDA when combined with one another in metastatic pancreatic adenocarcinoma. This arm will consist of gemcitabine 1000 mg/m2 IV day 1, 8 and 15 combined with nab-paclitaxel at 125 mg/m2 IV day 1, 8 and 15 every 28 days. Patients will be randomized equally to the two treatment arms. Primary objective is to assess progression-free survival (PFS). Toxicity assessment, response and overall survival are secondary endpoints. Statistical power is based on the comparison to historical control within each treatment arm. In particular, a sample size of 23 patients in each arm will have 84% power to differentiate the 3-month PFS of 30% (null hypothesis) versus 60% (alternative) based on a 2-sided test at a significance level of 0.05. There will be a lead-in phase to this trial for each treatment arm with a cohort size of 3 and a maximum of 6 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven newly diagnosed stage IV or stage IIIB non-squamous Non-small Cell Lung Cancer (NSCLC) - Recurrent advanced NSCLC will be allowed if they have never received chemotherapy for metastatic disease. - Prior adjuvant chemotherapy will be allowed, if recurrence occurred ≥ 6 months after last treatment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Washout period of 4 weeks for chemo/radiation/experimental agents
* Resolution of all toxicities to < grade 2 prior to starting treatment (excluding alopecia)
* Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE)
* Adequate hepatic, renal, and bone marrow functions
* Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment
* Negative serum or urine β-hCG pregnancy test at screening for patients of childbearing potential

Exclusion Criteria:

* Patient with New York Heart Association class III or IV heart failure
* Women of child bearing potential (WOCBP) are not currently pregnant or breast-feeding
* Co-existing malignancy or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma
* Previous anaphylactic or severe allergic reaction to paclitaxel and/or docetaxel will be excluded
* Grade ≥2 peripheral neuropathy at baseline assessment from any cause
* Symptomatic brain metastases will be excluded. Treated Brain metastases will be allowed that are neurologically stable.
* Patients with adenocarcinoma with activating EGFR mutation (exon 19 deletions / insertions, exon 21 point mutations) or EML4-ALK translocation are excluded unless they are ineligible for epidermal growth factor receptor (EGFR) or ALK targeting agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-15 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of first treatment until the date of first documented progression or date of death, which ever occurs first, assessed up to 60 months.
  To assess the progression-free survival (PFS) on patients with nab-paclitaxel and Gemcitabine at two different dose combinations and to compare the PFS to the historical data

SECONDARY OUTCOMES:
To explore differences in progression free survival (PFS) between two dose combinations of nab-paclitaxel with Gemcitabine in patients with advanced NSCLC. | From date of first treatment until the date of first documented progression or date of death, which ever occurs first, assessed up to 60 months.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Monga, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals - Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

REFERENCES:
- [Background] D'Addario G, Pintilie M, Leighl NB, Feld R, Cerny T, Shepherd FA. Platinum-based versus non-platinum-based chemotherapy in advanced non-small-cell lung cancer: a meta-analysis of the published literature. J Clin Oncol. 2005 May 1;23(13):2926-36. doi: 10.1200/JCO.2005.03.045. Epub 2005 Feb 22. PMID 15728229
- [Background] Jiang J, Liang X, Zhou X, Huang R, Chu Z, Zhan Q. Non-platinum doublets were as effective as platinum-based doublets for chemotherapy-naive advanced non-small-cell lung cancer in the era of third-generation agents. J Cancer Res Clin Oncol. 2013 Jan;139(1):25-38. doi: 10.1007/s00432-012-1294-z. Epub 2012 Aug 5. PMID 22864816
- [Background] Davidoff AJ, Tang M, Seal B, Edelman MJ. Chemotherapy and survival benefit in elderly patients with advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2191-7. doi: 10.1200/JCO.2009.25.4052. Epub 2010 Mar 29. PMID 20351329